CLINICAL TRIAL: NCT03149510
Title: A Patient-centered Mobile Intervention to Promote Self-management and Improve Patient Outcomes in Chronic Heart Failure
Brief Title: The Effects of Self-monitoring With a Mobile Application in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Todd M Koelling, MD, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00123222
Record Dates: First submitted 2017-04-20; First posted 2017-05-11 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure
Keywords: mobile application; mHealth
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application (Experimental): Participants will be using a mobile application, activity monitor and scale.
  Interventions: Behavioral: Mobile Application
- Control Group (No Intervention): Participants will receive standard of care.

INTERVENTIONS:
Behavioral: Mobile Application — Participants will use the mobile application daily to assess heart failure symptoms.
  Arms: Mobile Application

SUMMARY:
In the United States, about 40 percent of heart failure (HF) patients are readmitted within 1-year following their first admission for HF and hospitalization accounts for approximately 70 percent of the costs of HF management. As a result, the management of HF patients is evolving from the traditional model of face-to-face follow-up visits toward a proactive real-time technological model of assisting patients with monitoring and self-management while in the community. The investigators plan to test the impact of a mobile application on clinical outcomes in HF.

DETAILED DESCRIPTION:
HF patients with a reduced ejection fraction will be randomized to the mobile application versus placebo for 12 weeks. The mobile application will provide the participants with a reminder to perform self-monitoring, a health status indicator and heart failure education for self-management.

All participants will complete the Minnesota Living with Heart Failure Questionnaire and Self-Care Heart Failure Index. Hospital admissions and mortality will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* 45 years old or older
* Left ventricular ejection fraction </= 40% or an LVEF > 40% (with left atrial size >40mm or BNP > 200 pg/ml or NT-proBNP > 800 pg/ml)
* Admitted for acutely decompensated heart failure or recently discharged in the past 4 weeks.
* Smartphone (iOS or Android) with home wifi

Exclusion Criteria:

* Unstable coronary syndrome within 8 weeks (unstable angina, NSTEMI, STEMI)
* Primary valvular heart disease
* Known pericardial disease (Sarcoidosis, amyloidosis, rheumatoid arthritis, lupus)
* Uncorrected thyroid disease
* Advanced renal disease (dialysis or creatinine >4.0 mg/dL)
* End-stage HF (hospice candidate, home milrinone or dobutamine)
* Active cancer
* Pulmonary fibrosis
* Discharge to a setting other than home

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | Change from Baseline MLHFQ at Week 12
  MLHFQ is a quality of life questionnaire for heart failure.

SECONDARY OUTCOMES:
Self-Care Heart Failure Index (SCHFI) | Change from Baseline SCHFI at Week 12
  SCHFI is a survey of heart failure patient self-management.
Hospitalizations | Over 12 weeks
  Admission to the hospital while enrolled in the trial.
Mortality | Over 12 weeks
  Death while enrolled in the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Koelling, MD, Principal Investigator — University of Michigan Heart Failure Program
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorsch MP, Farris KB, Bleske BE, Koelling TM. A web application for self-monitoring improves symptoms in chronic systolic heart failure. Telemed J E Health. 2015 Apr;21(4):267-70. doi: 10.1089/tmj.2014.0095. Epub 2015 Feb 5. PMID 25654615
- [Background] Bleske BE, Dillman NO, Cornelius D, Ward JK, Burson SC, Diez HL, Pickworth KK, Bennett MS, Nicklas JM, Dorsch MP. Heart failure assessment at the community pharmacy level: a feasibility pilot study. J Am Pharm Assoc (2003). 2014 Nov-Dec;54(6):634-41. doi: 10.1331/JAPhA.2014.14039. PMID 25379983
- [Derived] Dorsch MP, Farris KB, Rowell BE, Hummel SL, Koelling TM. The Effects of the ManageHF4Life Mobile App on Patients With Chronic Heart Failure: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Dec 7;9(12):e26185. doi: 10.2196/26185. PMID 34878990